CLINICAL TRIAL: NCT07115927
Title: pReOperative Dostarlimab and Novel Therapies in EndOmetrial Cancer
Acronym: RODEO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/157607
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer
Keywords: Window of opportunity
MeSH Terms: conditions — Endometrial Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: Window of opportunity. This trial has been designed to run as a platform trial. Additional arms are in development.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Dostarlimab monotherapy (Experimental): Patients in the initial cohort will be treated with two doses of dostarlimab prior to surgery, receiving dostarlimab 500mg IV on day 1 and day 22.
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Arm 1: Patients in the initial cohort will be treated with two doses of dostarlimab prior to surgery, receiving dostarlimab 500mg IV on day 1 and day 22.

SUMMARY:
RODEO is a window of opportunity trial using dostarlimab in patients with newly diagnosed high-risk (stage 2-4) endometrial cancer who are suitable for primary surgery. Patients will receive 2 doses of dostarlimab (500mg IV day 1 and day 22) prior to surgery. The primary objective is to assess the pathological response rate to pre-operative dostarlimab and the secondary objectives are to assess the feasibility, toxicity, safety and efficacy of pre-operative dostarlimab.

DETAILED DESCRIPTION:
Background Endometrial cancer is the most common invasive gynaecological malignancy and its incidence is predicted to double by 2030. Surgery remains the most effective treatment modality to cure operable early-stage and high-risk cancers but despite the use of adjuvant therapies, a proportion of patients will relapse due to the presence of micrometastases that cannot be detected at the time of primary treatment. Immune checkpoint inhibitors have been evaluated in endometrial cancer, for example, the GARNET trial demonstrated the benefit of dostarlimab (anti-PD1) in women with relapsed/advanced endometrial cancer. Pre-operative immunotherapy is an evolving strategy that consists of administering an ICI, either as monotherapy or in combination before surgical resection in high-risk resectable disease, in the window between diagnosis and primary surgery

Aims RODEO is a proposed window trial using dostarlimab in patients with newly diagnosed high-risk (stage 2-4)endometrial cancer who are suitable for primary surgery. The primary objective is to assess the pathological response rate to pre-operative dostarlimab and the secondary objectives are to assess the feasibility, toxicity, safety and efficacy of pre-operative dostarlimab.

Methods Patients will receive 2 doses of dostarlimab (500mg IV day 1 and day 22) prior to surgery.

How the results of this research will be used. This trial will investigate the efficacy and safety of dostarlimab in this setting and multiple translational and clinical endpoints will be explored. It will provide a unique opportunity to study the immune microenvironment in treatment naïve tumours and help determine key mechanisms involved in the response and resistance to therapy, with the potential to develop biomarkers which may elucidate response beyond MMR status, so widening the potential benefit of this agent and assisting in future patient selection.

ELIGIBILITY:
1. Patient is at least 18 years of age.
2. Patient is able to provide informed consent and able to comply with treatment and follow up schedule.
3. Patients with surgically operable FIGO (2009) stage 3-4 endometrial cancer.
4. Must not have received any systemic anti-cancer treatment (including chemotherapy, hormonal therapy, immunotherapy, surgical intervention, radiotherapy) for the current diagnosis of endometrial cancer.
5. Histological diagnosis of advanced epithelial endometrial cancer (excluding carcinosarcoma).
6. CT or MRI proven disease (measurable or non-measurable).
7. Willing to provide tissue from archival diagnostic sample, a newly obtained core or excisional biopsy of a tumour lesion at screening and also collection of tissue during surgery.
8. Mismatch repair status must be known at time of enrolment. Patients can be screened based on local MMR/MSI testing results using immunohistochemistry (IHC), polymerase chain reaction (PCR), or next generation sequencing (NGS) performed in a certified local laboratory, i. MMR status must be assessed by immunohistochemistry (IHC) for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicates dMMR; dMMR may be determined locally.

   ii. MSI status as determined by polymerase chain reaction (PCR) or by tissue Next generation sequencing (NGS).

   Note: Patients who are known to have Lynch syndrome and have been found to carry a specific germline mutation in an MMR gene (MLH1, MSH2, MSH6, PMS2) and have dMMR or MSI-H in the tumour are eligible to participate.
9. Patient must have a negative serum pregnancy test within 24 hours prior to the date of the first dose of trial medication; unless they are of non-childbearing potential.

   Non-childbearing potential is defined as:

   i. ≥ 45 years of age and has not had menses for > 1 year. ii. Amenorrheic for < 2 years without a hysterectomy and oophorectomy and have a follicle-stimulating hormone (FSH) value in the postmenopausal range upon pre-trial evaluation.
10. Patients should have adequate bone marrow and laboratory functions defined as:

    * Absolute neutrophil count (ANC) ≥1.5×109/L
    * Haemoglobin ≥9 g/dL ≥5.6 mmol/L
    * Platelets ≥100×109/L
    * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5×ULN
    * Bilirubin ≤1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
    * For patients not taking warfarin: International normalized ratio (INR) <1.5 or prothrombin time (PT) <1.5×ULN and partial thromboplastin (PTT) <1.5×ULN. Patients taking warfarin may be included on a stable dose with a therapeutic INR <3.5.
    * Renal function parameters of GFR ≥30 mL/min/1.73m2 (institutional creatinine ≤1.5×ULN)
    * Albumin > 30
11. ECOG Performance Status 0 or 1.
12. Life expectancy of at least 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | At time of surgery
  To assess the pathological response rate to pre-operative treatment in patients with operable (FIGO (2009) stage 3-4) endometrial cancer

IPD SHARING:
Plan to Share IPD: No